CLINICAL TRIAL: NCT05897879
Title: Impact of Bacterial Expression and Immune Response in the Severity of Pertussis
Acronym: PERT-SEVEREII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Hôpital Necker-Enfants Malades (Other); Hospices Civils de Lyon (Other); Hopital Universitaire Robert-Debre (Other); Centre Hospitalier Intercommunal Creteil (Other); Nantes University Hospital (Other); Réseau ACTIV (Unknown); Hôpital Armand Trousseau (Other); CHR - Hôpital Roger Salengo (Unknown); Hôpital Nord - APHM (Unknown); Hôpital Louis Mourier (Other); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); Hôpital de la Timone (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-093; 2023-A00004-41 (Other: ID RCB)
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Bordetella Pertussis, Whooping Cough
Keywords: vaccination
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children between 0 and 15 years with suspected pertussis (Other)
  Interventions: Biological: Nasopharyngeal swab; Biological: Blood samples

INTERVENTIONS:
Biological: Nasopharyngeal swab — For hospitalized patients :
  Nasopharyngeal swab (1 aspiration or 2 swabs (1 in each nostril))
  For ambulatory patients :
  Deep nasal swab: 2 swabs (1 in each nostril), or 1 swab only for children for whom taking 2 swabs is complicated.
Biological: Blood samples — For hospitalized patients : 3 to 7.5 ml For ambulatory patients: Fingertip blood sampling

SUMMARY:
The resurgence of pertussis is associated with an evolutionary mechanism under the pressure of current acellular vaccines, with a possible impact on vaccine effectiveness and disease expression. Little is known about the mechanisms involved in the clinical variability of pertussis, including its most severe malignant form observed in infants (mortality between 50-80%). The main challenges are: (i) the lack of knowledge about the gene expression of B. pertussis strains currently circulating during human infection, incorporating evolutionary changes and vaccine-induced selective pressure; (ii) the poor understanding of the variability in clinical expression of pertussis, and (iii) the lack of biomarkers to predict disease severity or prognosis in infants.

An integrative strategy combining a clinical, microbiological, immunological and 'omic' approach from a prospective cohort of children with pertussis will be used to identify

1. 'in situ' expression profiles of B. pertussis genes and proteins incorporating recent evolutionary changes and
2. a systemic and respiratory immune signature in B. pertussis-infected children according to severity.

Results should furthermore serve as a prerequisite for the identification of severity biomarkers and new vaccine antigen candidates taking into account specific immune responses in infants.

DETAILED DESCRIPTION:
The study design is characterized by 4 work packages:

1. Collection of clinical data and biological samples (deep nasal swab, blood sample) from children with pertussis
2. Construction and validation of a microbial panel of 200 genes of interest (involved in virulence and/or potential vaccine antigens) for transcriptomic analysis
3. Transcriptomic study using the panel of interest of B. pertussis isolates from nasopharyngeal swabs preserved with an RNA stabilizer, using the Nanostring® technique
4. Study of the immune response during pertussis

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 0 and 15 years inclusive
* be suspected of having pertussis by the physician in charge, with the prescription of a diagnostic PCR (pertussis PCR, which may be a syndromic PCR, a PCR targeting IS481 and/or IS1001)
* be free of any pathology/treatment that may influence the immune response (autoimmune/inflammatory pathology or immune deficiency not listed above, hepatic insufficiency, taking immunosuppressive treatment (including taking oral corticosteroids with a dose ≥ 10 mg/d Prednisone equivalent for more than 15 days)
* Have received age-appropriate information and written assent or consent from their parents/legal guardians
* be affiliated with or benefiting from a social security plan

Exclusion Criteria:

* Patient with any pathology/treatment that may influence the immune response (autoimmune/inflammatory pathology or immune deficiency not listed above, hepatic failure, taking immunosuppressive therapy (including oral corticosteroids with dose ≥ 10 mg/d prednisone equivalent for more than 15 days)
* Use of antibiotics active against pertussis in the 24 hours preceding the sampling
* Delay between the result of the diagnostic sample (pertussis PCR) and the day of inclusion > 48 hours
* Patient's condition that, in the opinion of the physician, is incompatible with the expanded/additional sampling(s) required by the study
* Infant with a weight < 2.5 kg at the time of inclusion.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-11-16 (Estimated); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Measurement of expression level of Bp genes during infection by Nanostring transcriptomic analysis of Bp isolates from the nasopharynx of children with pertussis. | 3 years
  To identify in a standardized way the microbial "in situ" expression profiles of currently circulating Bp genes during infection in children ;
Measurement of plasma cytokine and chemokine concentrations by SIMOA digital ELISA | 3 years
  To determine systemic and respiratory immune responses in children during pertussis.
Phenotyping of immune cells by cytometry with a 20-color flow cytometry panel | 3 years
  To determine systemic and respiratory immune responses in children during pertussis.

SECONDARY OUTCOMES:
Measurement of expression level of Bp genes which is modified by recent gene developments related to vaccine pressure by Nanostring transcriptomic analysis of Bp isolates | 3 years
  List of microbial genes which expression is modified by recent genomic developments related to vaccine pressure
Measurement of high expression level of Bp genes in all clinical forms of pertussis by Nanostring transcriptomic analysis of Bp isolates | 3 years
  To identify new candidate Bp genes for a future protein vaccine
Measurement of expression level of Bp genes which is associated with severe pertussis by Nanostring transcriptomic analysis of Bp isolates | 3 years
  List of virulence genes differentially expressed during severe pertussis

CONTACTS AND LOCATIONS:
Overall Officials: Julie Toubiana, MD, Study Director — Institut Pasteur
Locations (14):
- France (14):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Louis Mourier, Colombes
  - Centre hospitalier intercommunal de Créteil, Créteil
  - Hôpital Roger Salengo, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital de la Timone Enfants, APHM, Marseille
  - Hôpital Nord, APHM, Marseille
  - CHU de Nantes, Nantes
  - CHU Armand Trousseau, Paris
  - Hopital Necker, Paris
  - Hôpital Robert Debré, Paris
  - CHU Rouen, Rouen
  - Réseau ACTIV, Saint-Maur-des-Fossés
  - CHU de Toulouse, Toulouse